CLINICAL TRIAL: NCT01473147
Title: Additional GLP-1 Analogue on CSII Treatment for Poorly Controlled Type 2 Diabetic Patients
Acronym: AGAC2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMRPG3A0911
Record Dates: First submitted 2011-11-14; First posted 2011-11-17 (Estimated); Last update posted 2013-07-30 (Estimated); Status verified 2011-11

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: GLP-1 analogue; CSII; insulin; type 2 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Exenatide; Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- GLP-1 (Active Comparator)
  Interventions: Drug: Exenatide
- Normal saline (Placebo Comparator)
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Exenatide — Exenatide 5 microgram bid sc.
  Other Names: Byetta
  Arms: GLP-1
Drug: Normal saline — Normal saline 2 u bid sc.
  Arms: Normal saline

SUMMARY:
Background: Continuous subcutaneous insulin infusion (CSII) has been demonstrated to be an effective clinical tool for intensive insulin therapy in Type 1 diabetic patients. Type 2 diabetes patients have been proved to have decreased of glucagon-like peptide-1 (GLP-1) levels. Injection of GLP-1 receptor agonists are associated with improved glycemic control. Nevertheless, the clinical effects and mechanisms are still unclear when additional supplement of GLP-1 analogue in cooperation with intensive CSII treatment for poorly controlled Type 2 diabetes patients. This study is designed to understand the complementary pharmacological effects of GLP-1 analogue on intensive CSII treatment.

Methods: Sixty poorly controlled Type 2 diabetes patients will be admitted to the ward for 6 days CSII intensive treatment. Following the normalization of blood glucose at first 3 days, the patients are randomly assigned with combined therapy with exenatide injection or saline for another 3 days. The clinical assessments of insulin requirement, insulin secretion, insulin resistance glycemic excursions and cytokines will perform immediately during or after the study.

DETAILED DESCRIPTION:
In the poorly controlled type 2 DM, insulin therapy is the treatment of choice to make sugar on target. Actually, however, the general control rate is not good and partially due to the complex etiology in type 2 DM. GLP-1 deficiency is the mostly emphasized in modern practice. In order to study the effect of GLP-1 analogue in insulinized type 2 DM patients, investigators have to optimize the insulin therapy in the first priority. Continuous subcutaneous insulin infusion (CSII) or insulin pump is a viable choice for patients with type 1 or type 2 DM who want close-to-physiologic insulin treatment. By means of the insulin pump therapy, standardized sugar control profile in type 2 DM patients could be achieved in a short time. Investigators can further evaluate the clinical response under GLP-1 analogue or not.

ELIGIBILITY:
Inclusion Criteria:

* Age > 20 years old
* DM diagnosed > 2 years
* HbA1c level of 8% to 12%
* Receiving insulin premixed insulin twice daily and total insulin daily dose > 0.6 u/kg/day

Exclusion Criteria:

* Severe comorbidity, including CHF, CVA, liver cirrhosis, COPD, Cushing's syndrome etc.
* Psychologic problems, including anxiety
* Incorporation, including personal and familial factors

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2011-10; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Mean amplitude of glycaemic excursions (MAGE) | During 6-day treatment course

SECONDARY OUTCOMES:
homeostasis model assessment(HOMA) | During 6-day treatment course

CONTACTS AND LOCATIONS:
Overall Officials: CHIA-HUNG LIN, M.D., Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan